CLINICAL TRIAL: NCT03732716
Title: The Relationship Between Sarcopenia and Orthostatic Hypotension
Brief Title: Sarcopenia and Orthostatic Hypotension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kudret Keskin, Principle Investigator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2052
Record Dates: First submitted 2018-09-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Orthostatic Hypotension; Sarcopenia
Keywords: blood pressure; elderly; sarcopenia; fall
MeSH Terms: conditions — Hypotension, Orthostatic; Sarcopenia | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly with sarcopenia: 50 patients aged 75 or older with sarcopenia Intervention: Each patient's supine and standing blood pressures will be measured.
  Interventions: Diagnostic Test: blood pressure measurement
- Elderly without sarcopenia: 50 patients aged 75 or older without sarcopenia Intervention: Each patient's supine and standing blood pressures will be measured.
  Interventions: Diagnostic Test: blood pressure measurement

INTERVENTIONS:
Diagnostic Test: blood pressure measurement — Intervention: Each patient's supine and standing blood pressure measurements will be recorded

SUMMARY:
Elderly patients generally have a tendency for having sarcopenia which refers to muscle loss that may be related to many factors. These patients also have a tendency to falls and injuries. Whether elderly sarcopenic patients have abrupt blood pressure drops upon standing remains unknown. Therefore, in this study, we sought to determine the incidence of orthostatic hypotension in sarcopenic elderly patients and compare it with elderly patients with no sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years or older

Exclusion Criteria:

* Pace-maker
* End stage renal insufficiency
* End stage malignancy
* Dehydration
* Severe anemia ( Hgb < 8 gr/dl)
* Acute infection
* Marked edema
* Neurodegenerative disease

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients ( 75 or older) with and without sarcopenia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | 0-3 minutes
  All blood pressure measurements will be performed in the morning after an eight-hour fasting. After 5-minute rest, the first blood pressure measurement will be taken when the patients are supine. Later, three more consecutive measurements will be recorded when the patients stand up each being one-minute apart. All measurements will be performed using a fully automated sphygmomanometer that is attached with the correctly sized cuff matching to the patients' upper arm circumference. OH is defined as a decrease in systolic blood pressure of 20 mm Hg or a decrease in diastolic blood pressure of 10 mm Hg within 3 minutes of standing. The accompanying symptoms such as dizziness, unable to maintain balance, blurred vision will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Orta Kılıçkesmez, Prof, Study Director — Şişli Hamidiye Etfal Education and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Education and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Hashimoto Y, Kaji A, Sakai R, Hamaguchi M, Okada H, Ushigome E, Asano M, Yamazaki M, Fukui M. Sarcopenia is associated with blood pressure variability in older patients with type 2 diabetes: A cross-sectional study of the KAMOGAWA-DM cohort study. Geriatr Gerontol Int. 2018 Sep;18(9):1345-1349. doi: 10.1111/ggi.13487. Epub 2018 Jul 24. PMID 30039599